CLINICAL TRIAL: NCT01031082
Title: Identification and Characterization of the Bacteria Causing Acute Otitis Media (AOM) Episodes in HIV-positive and HIV-negative Children in South Africa
Brief Title: Study to Identify and Characterize Bacteria Causing Acute Otitis Media in South African Children
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Other Study IDs: 112135
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Last update posted 2010-05-24 (Estimated); Status verified 2010-05

CONDITIONS: Acute Otitis Media
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Middle ear fluid, nasopharyngeal aspirate and urine.

GROUPS / COHORTS (2):
- HIV-negative Group: This group is sub-divided into two sub-groups. One sub-group includes HIV-negative/ presumed negative subjects with a new episode of acute otitis media who have not yet received antibiotic therapy for the episode and the other sub-group includes HIV-negative/ presumed negative subjects with treatment failure who have had a diagnosis of acute otitis media and showed no clinical improvement within 48-72 hours of antibiotic treatment.
  Interventions: Procedure: Middle ear fluid, nasopharyngeal aspirate and urine sample.
- HIV-positive Group: This group is sub-divided into two sub-groups. One sub-group includes HIV-positive subjects with a new episode of acute otitis media who have not yet received antibiotic therapy for the episode and the other sub-group includes HIV-positive subjects with treatment failure who have had a diagnosis of acute otitis media and showed no clinical improvement within 48-72 hours of antibiotic treatment.
  Interventions: Procedure: Middle ear fluid, nasopharyngeal aspirate and urine sample.

INTERVENTIONS:
Procedure: Middle ear fluid, nasopharyngeal aspirate and urine sample. — Middle ear fluid, nasopharyngeal aspirate and urine sample collection.

SUMMARY:
The purpose of this study is to identify and characterize the bacteria causing acute otitis media episode in HIV-positive and HIV-negative children (>=3 months to <5 years) in South Africa. Middle ear fluid sampling either by tympanocentesis or by careful sampling of spontaneous otorrhoea will be done; nasopharyngeal aspirate and urine sample will also be collected from the subjects.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for all subjects:

* Age: >= 3 months and < 5 years at the time of enrolment.
* Signs, symptoms, and conditions:
* One of the functional or general signs of otalgia,, conjunctivitis, fever and either
* Paradise's criteria or
* Spontaneous otorrhoea of less than 24 hours.
* Subject will be included as a treatment failure case.
* Written informed consent obtained from parent or guardian prior to study start.

Inclusion criteria for HIV-positive subjects:

* Documented HIV-positive status as given in subject's medical records. or
* Subjects referred from paediatric HIV clinic.

Inclusion criteria for HIV-negative subjects (including presumed negative children)

* Children who have been tested HIV-negative.
* Children whose mothers volunteer to have tested HIV-negative whilst pregnant with the index case and the child is free to any World Health Organization Grade II stigmata of HIV/acquired immunodeficiency syndrome.
* Children who do not fulfil the World Health Organization staging for HIV infection / immunosuppression.

Exclusion Criteria:

* Hospitalised during the diagnosis of acute otitis media or during treatment.
* Otitis externa or otitis media with effusion.
* Presence of a transtympanic aerator.
* Systemic antibiotic treatment received for a disease other than acute otitis media in the 72 hours prior to enrolment.
* Receiving antimicrobial prophylaxis for recurrent acute otitis media but excluding cotrimoxazole or isoniazid prophylaxis in HIV exposed children.
* Provision of antibiotic by paediatrician/ENT specialist at the enrolment visit prior to the sampling of the middle ear fluid or spontaneous Otorrhoea.
* Children on antibiotics for acute otitis media who are clinically improving.

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged >= 3 months and < 5 years seeking healthcare for the treatment of acute otitis media.
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of bacterial pathogens isolated from middle ear fluid samples in HIV-positive and HIV-negative subjects.

SECONDARY OUTCOMES:
Occurrence of bacterial serotypes.
Antimicrobial susceptibility of different bacteria isolated from middle ear fluid samples as assessed by standard microbiological techniques.
Occurrence of treatment failure of acute otitis media and of recurrent acute otitis media.
Occurrence of spontaneous otorrhoea.
Occurrence of bacteria in acute otitis media cases with treatment failure and in new acute otitis media cases without treatment therapy.
Occurrence of bacteria in acute otitis media cases vaccinated with a pneumococcal vaccine.
Frequency of concurrent respiratory viral infection coinciding with the episode of acute otitis media.
The comparison of above endpoints in HIV-positive and HIV-negative subjects.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Soweto, Gauteng, South Africa

REFERENCES:
- [Derived] Madhi SA, Govender N, Dayal K, Devadiga R, Van Dyke MK, van Niekerk N, Cutland CL, Adrian PV, Nunes MC. Bacterial and Respiratory Viral Interactions in the Etiology of Acute Otitis Media in HIV-infected and HIV-uninfected South African Children. Pediatr Infect Dis J. 2015 Jul;34(7):753-60. doi: 10.1097/INF.0000000000000733. PMID 25923426